CLINICAL TRIAL: NCT07172698
Title: Effects of a Multicomponent Protocol With Emphasis on Muscle Power Training on Bradykinesia in Individuals With Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Fernanda Cechetti, Professor, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FUHSPortoAlegre_Minotto_Amado
Record Dates: First submitted 2025-07-28; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G1 - traditional multicomponent training (Experimental): Group 1 will perform an exercise protocol that includes warm-up, mobility, muscle strength, and flexibility
  Interventions: Other: traditional multicomponent training
- G2 - multicomponent training with an emphasis on muscle power (Experimental): Group 2 will perform the same exercise protocol, with the caveat that, whenever feasible, exercises will be executed in the muscle power modality (at the highest possible speed). This latter training is characterized by a lower number of repetitions and a higher movement speed, guided by the therapists assisting. The progression of muscle power exercises will occur at 35%, 40%, 45%, 50%, 55%, and 60% of 1RM over the 12 weeks, distributed in 2 sets of 6 to 8 repetitions, with rest times of 60 to 120 seconds.
  Interventions: Other: multicomponent training with an emphasis on muscle power

INTERVENTIONS:
Other: multicomponent training with an emphasis on muscle power — Group 1 will perform an exercise protocol that includes warm-up, mobility, muscle strength, and flexibility. Group 2 will perform the same exercise protocol, with the caveat that, whenever feasible, exercises will be executed in the muscle power modality (at the highest possible speed). This latter training is characterized by a lower number of repetitions and a higher movement speed, guided by the therapists assisting. The progression of muscle power exercises will occur at 35%, 40%, 45%, 50%, 55%, and 60% of 1RM over the 12 weeks, distributed in 2 sets of 6 to 8 repetitions, with rest times of 60 to 120 seconds.
  Arms: G2 - multicomponent training with an emphasis on muscle power
Other: traditional multicomponent training — Group 1 will perform an exercise protocol that includes warm-up, mobility, muscle strength, and flexibility
  Arms: G1 - traditional multicomponent training

SUMMARY:
Parkinson's disease (PD) is a chronic progressive neurological disorder that involves both motor and non-motor symptoms, culminating in functional decline and disability. One of the main symptoms of PD is bradykinesia and its deleterious effect on functionality. Muscle weakness has also been reported as an important symptom of PD, and muscle power may be even more affected and related to these symptoms. Typical conventional physical therapy treatment includes mobility exercises, strength training, gait training, and balance training, and it presents numerous benefits associated with the reduction of motor symptoms of PD. Physical therapy with power training has also been studied as an alternative to improve the ability to perform activities of daily living in other populations. However, the literature that includes power training in physiotherapeutic approaches for people with PD is scarce. Power training may minimize the problems arising from changes in motor function in older adults with PD; however, there is still a lack of evidence using this modality in the different subtypes of the disease. Knowing that motor function is associated with functional capacity and disease severity, physical therapy becomes an important treatment resource with exercises to improve muscle power. Therefore, the objective of this study is to investigate the effect of a multicomponent protocol with an emphasis on muscle power training concerning bradykinesia in individuals with rigid-akinetic type PD. A Randomized Clinical Trial will be conducted, in which individuals diagnosed with Parkinson's disease, rigid-akinetic type, classified from 1 to 3 on the Hoehn and Yahr Scale, aged between 50 and 85 years, and who sign the Informed Consent Form will participate. The individuals will be randomized into two treatment groups: G1 - traditional multicomponent training, and G2 - multicomponent training with an emphasis on muscle power. Assessments will be conducted at four time points for all participants: before (T0), during (T1 - 6 weeks), immediately after intervention (T3 - 12 weeks), and follow-up (T4 - 16 weeks). The assessments will consist of the analysis of: 1) motor function through the adapted Unified Parkinson's Disease Rating Scale (UPDRS III) (bradykinesia as the primary outcome); 2) mobility of the posterior chain of the trunk and lower limbs using the Wells Bench; 3) body composition by Dual-Energy X-ray Absorptiometry (DXA); 4) rigidity of the leg extensor muscles assessed by ultrasound elastography; 5) muscle power of knee extensors using a linear potentiometer (Peak Power, CEFISE); 6) functional capacity through the Vertical Jump - CMJ and the Sit-to-Stand Five Times Test (TSLCV); and 7) postural assessment using the NeuroPostureApp. Treatment sessions will occur twice a week for 12 weeks, lasting 60 minutes each, totaling 24 sessions for each intervention. Group 1 will perform an exercise protocol that includes warm-up, mobility, muscle strength, and flexibility. Group 2 will perform the same exercise protocol, with the caveat that, whenever feasible, exercises will be executed in the muscle power modality (at the highest possible speed). This latter training is characterized by a lower number of repetitions and a higher movement speed, guided by the therapists assisting. The progression of muscle power exercises will occur at 35%, 40%, 45%, 50%, 55%, and 60% of 1RM over the 12 weeks, distributed in 2 sets of 6 to 8 repetitions, with rest times of 60 to 120 seconds.

ELIGIBILITY:
Inclusion Criteria:

To be included in the research, individuals must:

* be Diagnosed with Parkinson's disease and classified as 1 to 3 on the Hoehn and Yahr Scale;
* Present rigid akinetic PD;
* Be Aged between 50 and 85 years;
* Achieve a minimum score of 21 points on the Montreal Cognitive Assessment (MoCa);
* Sign the Informed Consent Form (ICF)

Exclusion Criteria:

Individuals will be excluded from this study if they present:

* Previous associated neurological diseases;
* Vestibular system disorders;
* Change in the pattern of levodopa use during the study;
* Severe heart disease;
* Uncontrolled arterial hypertension;
* Previous spinal surgeries;
* Tumors or infection of the spinal column;
* Inflammatory diseases of the spinal column;

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Bradykinesia | Baseline, 6 weeks, end of intervention (12 weeks) and follow-up (16weeks)
  The objective of this study is to investigate the effect of a multicomponent protocol with an emphasis on muscle power training concerning bradykinesia in individuals with rigid-akinetic type PD. This outcome will be measured using the UPDRS (Unified Parkinson's Disease Rating Scale) Part III.

SECONDARY OUTCOMES:
Mobility of the posterior chain of the trunk and lower limbs | Baseline, 6 weeks, end of intervention (12 weeks) and follow-up (16weeks)
  Sit and Reach (SA) Test on the Wells Bench This tool allows the assessment of the amplitude and flexibility of the back of the trunk and lower limbs. To perform the test, the Wells bench is used, where individuals are instructed to sit with their feet in full contact with the front of the bench and their lower limbs with their hips flexed and their knees extended. The subjects are instructed to perform a trunk flexion together with a forced exhalation and to move the bench scale as far as they can. This procedure is performed three times and immediately noted by the evaluator; the value obtained in each attempt is expressed in centimeters, and the best one is selected.
Body composition by Dual-Energy X-ray Absorptiometry (DXA) | Baseline, 6 weeks, end of intervention (12 weeks) and follow-up (16weeks)
  Dual-energy X-ray absorptiometry (DXA) is a method used to assess body composition. DXA is one of the most accurate and consistent techniques for evaluating body composition, particularly in quantifying fat mass, lean mass, and bone mineral density (SANTOS et al., 2022).
  The composition of the dominant lower limb thigh of the participant will be estimated using dual-energy X-ray absorptiometry with a Lunar Prodigy Advance device (GE Healthcare, Chicago, IL, USA). According to the manufacturer's recommendations, prior to scanning, participants will be asked to remove all removable metal-containing objects (e.g., jewelry, glasses, clothing with buttons or zippers). Scans will be performed with participants lying in a supine position along the longitudinal axis of the scanner table's centerline. The feet will be tied together to immobilize the legs, while the hands will be placed in a prone position within the scanning region. All assessments will be conducted by the same examiner. DXA
Rigidity of the leg extensor muscles assessed by ultrasound elastography | Baseline, 6 weeks, end of intervention (12 weeks) and follow-up (16weeks)
  To analyze stiffness by elastography, an ultrasound device (Nemio XG, Toshiba, Japan), tape measure, dermographic pen, and water-soluble gel will be used.
  Muscle thickness (MT, mm) and subcutaneous fat thickness (SFT, mm) of the vastus lateralis, rectus femoris, and vastus intermedius muscles of the right limb will be measured using B-mode imaging using an ultrasound device (Nemio XG, Toshiba, Japan) with a 7.5 MHz linear probe (38 mm depth, 90 dB gain).
  Before imaging begins, to allow for the distribution of body fluids, participants will lie supine for 5 minutes with their lower limbs extended and relaxed, and must remain in this position throughout the assessment. A water-soluble gel, which promotes acoustic contact without applying pressure to the skin, will be applied to the assessment site, and the transducer will be positioned perpendicular to the assessed muscles.
Muscle power of knee extensors using a linear potentiometer (Peak Power, CEFISE) | Baseline, 6 weeks, end of intervention (12 weeks) and follow-up (16weeks)
  The linear potentiometer (Peak Power, CEFISE) consists of an electronic system interfaced to software that measures the displacement speed of any body within a range of up to 2.5 meters. The speed is measured by a precision stopwatch connected to a wire that can be attached to the dumbbell or weight column of the equipment. The use of a linear encoder to assess power has been proven to be safe in people with Parkinson's disease (BONDE-JENSEN et al., 2024). Muscle power will be assessed on the KONNEN GYM® knee machine.
Functional capacity through the Vertical Jump - CMJ | Baseline, 6 weeks, end of intervention (12 weeks) and follow-up (16weeks)
  The analysis of the vertical jump allows the collection of several metrics (flight time, exit speed and joint angle). Based on these measurements, it is possible to estimate other significant values such as muscle power of the lower limbs and jump height (LOTURCO et al., 2017). A verification of the complete movement can be performed (separation of each stage and the influence of these stages on the performance of the individuals) or, in a more simplified way, only the height of the jump can be considered. This estimate is generally made based on the flight time and assuming constant acceleration of the individual's center of mass (CONCEIÇÃO et al., 2022). To obtain these metrics, we will use a force platform (Cefise - Jump, System Pro, software version 1.0, Brazil).
  The signal will be captured at a frequency of 1000 Hz and the force platform will be calibrated before all tests according to the manufacturer's instructions.
Sit-to-Stand Five Times Test | Baseline, 6 weeks, end of intervention (12 weeks) and follow-up (16weeks)
  The TSLCV can be used to assess functional mobility, including risk of falling, balance and measurement of lower limb strength in people with Parkinson's.
  The individual begins the test sitting in a chair without arms and is instructed to stand with arms crossed over the chest; with full extension of the hips and knees, returning to a sitting position with the back supported by the vertical back of the chair. It should be repeated 5 times sequentially and without interruption; recording the total time taken to perform the test. A risk of falling is suggested when the individual performs the test for more than 16 seconds (DUNCAN, 2011).
Postural assessment using the NeuroPostureApp | Baseline, 6 weeks, end of intervention (12 weeks) and follow-up (16weeks)
  The postural assessment will be performed using the NeuroPostureApp application, which is available free of charge in full (http://www.neuroimaging.uni-kiel.de/NeuroPostureApp). This instrument allows you to use a photo in a lateral view to assess camptocormia using the reference points (lateral malleolus, L5 and C7) (SCHLENSTEDT, 2020).

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil